CLINICAL TRIAL: NCT05328388
Title: A 12-week Clinical Study to Evaluate the Efficacy of Oral Lycomato Supplement on Skin Health and Appearance in Healthy Participants.
Brief Title: A Study to Evaluate the Effect of Lycomato on Skin Attributes in Healthy Participants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRSI-E-ES-094155-01-10-21
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Skin
MeSH Terms: interventions — Lycopene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lycomato (Experimental): Lycomato soft gel
  Interventions: Dietary Supplement: Lycomato

INTERVENTIONS:
Dietary Supplement: Lycomato — Lycomato sof gels

SUMMARY:
The study will be performed with oral gels, with up to 55 study subjects who meet the inclusion and non-inclusion criteria required. Study subjects will be instructed to use the products during 12 weeks and they will be assessed and supervised throughout the study by clinic technicians, in order to check for possible adverse events. Efficacy documentation through digital photography, instrumental measurements with the devices Cutometer® MPA 580 and Tewameter®, image acquisition with Visia-CA® as well as self-assessment through questionnaires will be carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Females in good general health, and between ages of 35 and 55 years old, inclusive at enrollment;
2. 50 subjects: 20 Caucasians + 10 Asians + 10 African Americans + 10 Latinos;
3. All Fitzpatrick skin types being II, III and IV for Caucasian/Asian;
4. Subjects to have Glogau skin classification of photoaging, Type 2;
5. Subjects with baseline signs of facial skin aging as conformed by visual expert grading of photographs

Exclusion Criteria:

1. Subjects participating in any other clinical studies;
2. Subjects that underwent beauty injections/ deep pealing/ cosmetic surgery/ tanning- for 3 months before study starts and for all the study duration.
3. Subjects having an acute or chronic disease or medical condition, including dermatological problems, which could put her at risk in the opinion of the Principal Investigator or compromise study outcomes. Typical uncontrolled chronic or serious diseases and conditions which would prevent participation in any clinical trial are cancer, AIDS, diabetes (insulin dependent), renal impairment, mental illness, drug/alcohol addiction;
4. Unreliable or unlikely to be available for the duration of the study;
5. History of allergic reactions, skin sensitization and/or known allergies to cosmetic ingredients, toiletries, sunscreens, etc.;
6. Immunocompromised subjects

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Expert clinical grading of efficacy attributes | 12 weeks
  Visual assessments will be performed by the expert grader using a 10-point ordinal scale on the face.

CONTACTS AND LOCATIONS:
Locations (1):
- Media Lab Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No